CLINICAL TRIAL: NCT02805218
Title: The Multi-center,Open-label,Single Arm Clinical Trial of Efficacy and Safety of PEG-rhG-CSF in Patients With Lymphoma Receiving Chemotherapy
Brief Title: PEG-rhG-CSF in Patients With Lymphoma Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-PGC-IV-02-1
Record Dates: First submitted 2016-06-13; First posted 2016-06-17 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim

ARMS (1):
- PEG-rhG-CSF (Experimental): patients received a single dose of 100 ug/kg of PEG-rhG-CSF(pegfilgrastim), on the basis of actual body weight, as a single subcutaneous injection on day 3 after chemotherapy
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF
  Other Names: pegfilgrastim

SUMMARY:
The purpose of this study is to estimate the safety and efficacy of PEG-rhG-CSF in patients with lymphoma receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥ 18 years
* diagnosis of lymphoma(Hodgkin's lymphoma and non-Hodgkin's lymphoma) patients
* Karnofsky Performance Status Z70
* life expectancy of at least 8 months
* normal white blood cell count and platelet count
* Written informed consent are acquired

Exclusion Criteria:

* uncontrolled infection
* pregnancy
* Have accepted any other anti-tumor drug within 4 weeks before anticipated the study
* Other situations that investigators consider as contra-indication for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2013-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
The occurrence rate of adverse event | up to 30 days after the patient study completion
The severity of adverse event | up to 30 days after the patient study completion

SECONDARY OUTCOMES:
the occurrence rate of grade III/ IV neutropenia during chemotherapy cycles | through the study completion,an average of 5 months